CLINICAL TRIAL: NCT06451575
Title: Thrombophilia and Tendency to Thrombosis in Behçet's Disease
Brief Title: Thrombophilia and Thrombosis in Behçet's Disease
Status: Recruiting | Type: Observational
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Erdal Pala, assistant professor doctor, Ataturk University
Other Study IDs: 30.03.2023/219
Record Dates: First submitted 2024-05-23; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Behçet Disease
Keywords: thrombosis; thrombophilia; Behcet's disease
MeSH Terms: conditions — Behcet Syndrome; Thrombosis; Thrombophilia | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA isolation will be performed with DNA isolation kit from peripheral blood in EDTA tube taken from patients during routine examinations. DNA samples will be stored at -20 degrees centigrade until the time of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases with Behcet's disease: Behcet's disease
  Interventions: Diagnostic Test: Blood collection
- healthy individuals: Healthy control group
  Interventions: Diagnostic Test: Blood collection

INTERVENTIONS:
Diagnostic Test: Blood collection — Blood collection

SUMMARY:
Behçet's disease (BD) is a systemic vasculitis of unknown cause, affecting mainly young adults. Vasculopathy has been reported in 16.8-51.5% of cases. Genetic, infectious factors, environmental factors, presence of autoantibodies, endothelial pathologies and hypercoagulability are responsible for the etiopathogenesis of BD. The main involvements responsible for morbidity and mortality in Behçet's disease are ocular, major cardiovascular and neurological involvements. Although there is an increased thrombotic risk in the etiopathogenesis of Behçet's disease, the cellular and molecular mechanisms are not fully understood. Although endothelial dysfunction due to inflammation has been shown to be the primary cause of vascular damage in Behçet's disease, some clinical evidence suggests that hypercoagulable states also contribute to thrombosis. The most common form of vascular involvement in Behçet's disease is deep vein thrombosis in the lower extremities. Arterial occlusion mostly affects the subclavian and pulmonary arteries. Although arterial involvement is rarer than venous involvement in Behçet's disease, morbidity and mortality are higher than venous involvement.

Although an increased thrombotic risk is mentioned in the etiopathogenesis of Behçet's disease, it is still controversial whether vasculitis or susceptibility to hypercoagulability plays a role in the pathogenesis of venous thrombosis. In addition, there are very few studies in the literature in which all thrombophilic parameters were analysed. Again, there is no recent study on this subject. The aim of our study is to determine the risk of hypercoagulability in Behçet's disease patients with vascular involvement, which has a highly mortal course.

DETAILED DESCRIPTION:
The study was planned as a prospective case control study. The study will be conducted on 100 Behçet's patients aged 18-70 years who were diagnosed with Behçet's disease according to the International Behçet's diagnostic criteria and 100 healthy controls similar in age and gender who applied to Atatürk University Faculty of Medicine Dermatology outpatient clinic between June 2023 and September 2024. Routine clinical evaluations of all patients will be performed. Demographic characteristics (age, gender), clinical features of the disease and medications used will be recorded. Patients will be included in the study after the relevant department consultations for system involvement. Skin and mucous membrane findings seen in the last 1 month will be recorded. Blood samples will be taken from all participants and analysed in the Genetics laboratory of our hospital. DNA isolation will be performed with DNA isolation kit from peripheral blood in EDTA tube taken from patients during routine examinations. DNA samples will be stored at -20 degrees Celsius until the time of the study. After collecting the targeted number of samples, Factor II G20210A, Factor V Leiden G1691A, MTHFR (Methylene Tetra Hydro Folate Reductase) C677T, MTHFR A1298C, Factor XIII V34L, PAI (Plasminogen Activator Inhibitor-1) 4G/5G SNP (single nucleotide polymorphisms) analyses will be performed with the thrombophilia panel kit. This analysis will be performed by fragment analysis method on the ABI 3130 Genetic analyser device in the Medical Genetics Laboratory. Firstly, PCR study will be performed with the thrombophilia panel kit, the plate with patient DNA will be loaded into the capillary electrophoresis device and the analyses will be interpreted and finalised with GeneMapper software.

ELIGIBILITY:
Inclusion Criteria:

1. 18-70 years old
2. Patients who fulfil the international diagnostic criteria for Behçet's disease
3. Those who accepted the consent form

Exclusion Criteria:

1. Those under 18 years of age
2. accompanied by another inflammatory dermatological disease
3. Pregnancy and breastfeeding
4. Those who use drugs that increase the tendency to thrombosis -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 patients with Behçet's disease aged 18-70 years and 100 age- and sex-matched healthy controls
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Faktor II G20210A kit | 15 months
  Faktor II G20210A at 200 participants
Faktor V Leiden kit | 15 months
  Faktor V Leiden at 200 participants
G1691A kit | 15 months
  G1691A at 200 participants
MTHFR (Methylene Tetra Hydro Folate Reductase) kit | 15 months
  MTHFR (Methylene Tetra Hydro Folate Reductase) at 200 participants
C677T kit | 15 months
  C677T at 200 participants
Factor XIII kit | 15 months
  Factor XIII at 200 participants
With DNA isolation kit | 15 months
  PAI (Plasminogen Activator Inhibitor-1) at 200 participants

CONTACTS AND LOCATIONS:
Overall Officials: ERDAL PALA, Principal Investigator — Ataturk University
Locations (1):
- Erdal Pala, Erzurum, Üniversite Mahallesi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No